CLINICAL TRIAL: NCT03283540
Title: The Short Term Implications of Transanal Total Mesorectal Excision (TaTME) for Rectal Cancer on Anal Physiology and Fecal Incontinence
Brief Title: Transanal Total Mesorectal Excision for Rectal Cancer on Anal Physiology + Fecal Incontinence
Status: Active, not recruiting | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE6217
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Rectal Cancer
Keywords: Low Anterior Resection
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Surgical specimen will be evaluated by a pathologist as part of the standard of care for the quality of resection and TME plane assessment.
  Resections will be categorized as follows: R0-all gross disease resected by enblocresection with margins histologically free of disease; R1-all gross disease resected byenblocresection with margins histologically positive for disease; and R2-residual gross disease remains unresected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TaTME: Trans-anal Total Mesorectal Excision (TaTME) is the visualization and dissection of the rectum located deep in the pelvis. In it, a trans-anal port is inserted for the duration of the surgery. Multiple surgical tools are then introduced through the port and the rectum is resected from down-to-up under direct visualization.
  Interventions: Procedure: TaTME
- abdominal TME: Total Mesorectal Excision involves resecting the rectum along with its surrounding Mesorectal plane. If the anal sphincter is spared, this surgery is named Low Anterior resection (LAR) for rectal cancer. Traditionally, TME dissection in LAR is performed through open or laparoscopic incisions(s) made in the abdominal wall. Mobilization of the splenic flexure along with sigmoid dissection follows. Lastly, the rectum is dissected in accordance with TME principles from above. This "up-to-down" approach is known as abdominal TME.
  Interventions: Procedure: TME

INTERVENTIONS:
Procedure: TaTME — Low anterior resection of the rectum entails a sharp dissection circumferentially around the mesorectum in an avascular plane between the visceral and parietal layers of the endopelvic fascia in what is known as Total Mesorectal Excision. This dissection can be achieved transanally starting down in the pelvis and going up in what is known as Transanal Total Mesorectal Excision
  Other Names: Trans-anal Total Mesorectal Excision
  Groups: TaTME
Procedure: TME — Low anterior resection of the rectum entails a sharp dissection circumferentially around the mesorectum in an avascular plane between the visceral and parietal layers of the endopelvic fascia in what is known as Total Mesorectal Excision. This surgery can also be done via an up-to-down approach beginning high in the abdomen and going low in the pelvis to achieve dissection around the mesorectum.
  Other Names: Total Mesorectal Excision
  Groups: abdominal TME

SUMMARY:
Low Anterior Resection (LAR) surgery can be done using various techniques. The traditional technique for performing the surgery is through one or multiple incision(s) in the muscular wall of the abdomen. This will allow the surgeon to gain access to inside the belly (Abdominal cavity). The surgeon will start from above and go down until reaching the rectum located low in the pelvis. The surgeon will then cut out the rectum along with some of the tissue surrounding it and reconnect the bowel.

An alternative new approach to perform Low Anterior Resection is called the Trans-anal approach. In this technique, a tube containing special surgical tools is introduced through the anus (back passage), while the patient is asleep. These tools are used to free the rectum up from its surroundings so that it can be removed.

Taking out the rectum via the opening of the anus (Trans-anal) is a relatively new surgical approach. This new technique enables the surgeon to better see deep in the pelvis which makes it easier to remove the rectum and its surrounding outer tissues while protecting other important nerves and organs located in the pelvis. However, it also involves inserting a tube through the opening of the anus to perform the rectal dissection. The alternative traditional way of doing the operation does not involve inserting such a tube because the access to the pelvis and rectum is gained from above through incision(s) in the abdominal wall.

The anal sphincter is the medical name for the muscle layers surrounding the opening of the anus. The anal sphincter functions as a seal that can be opened to discharge body waste and allow the passage of stool. A damage to the anal sphincter can result in inability to fully control bowel movements, causing stool (feces) to leak unexpectedly. Because the Trans-anal approach involves inserting a tube through the opening of the anus for the duration of the surgery, this can lead to a certain degree of stretch and damage to the anal sphincter muscles.

The main aim of this study is to compare the effect of the these two possible approaches to perform "Low Anterior Resection" operation on the muscles of the anal sphincter and whether they are associated with stool seepage from the anus after the operation.

Whether the patient is receiving the traditional or trans-anal approach is not related to the subject's participation in the study and is decided by the treating surgeon based on medical and surgical reasoning.

DETAILED DESCRIPTION:
Primary Objective To evaluate effect of TaTME on anal sphincter via anorectal functional studies and anorectal ultrasound administered post- and preoperatively.

Secondary Objective(s) To evaluate the effect of TaTME on fecal incontinence, quality of life, and LARS utilizing validated questionnaires administered to patients preoperatively and during postoperative follow-up.

Study Design This is a prospective two-arm cohort study. The study will include patients already undergoing the standard-of-care, low anterior resection (LAR) for middle to low rectal cancers. Low anterior resection of the rectum entails a sharp dissection circumferentially around the mesorectum in an avascular plane between the visceral and parietal layers of the endopelvic fascia in what is known as Total Mesorectal Excision (TME). This dissection can be achieved transanally starting down in the pelvis and going up in what is known as Transanal Total Mesorectal Excision- (TaTME). It can also be done via an up-to-down approach beginning high in the abdomen and going low in the pelvis to achieve dissection around the mesorectum. Access in the latter is achieved via laparoscopic or open abdominal incisions with minimal anal sphincter dilation. In addition, the level of coloanal anastomosis performed is potentially higher from the anal sphincter in comparison to TaTME. TaTME on the other hand, involves introducing a special port (gelpoint path) transanally to perform the TME dissection. In order to better evaluate the effect of TaTME on anal sphincter, it is quintessential to include a control group with minimal anal sphincter manipulation, thus the conventional abdominal (open or laparoscopic) TME group will serve as a control.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically confirmed Rectal Adenocarcinoma.
* Subjects must have Rectal Adenocarcinoma located up to 10 cm from the anal verge measured by preoperative MRI, proctoscopy, or digital rectal examination.
* Subjects must have treated with Transanal total mesorectal excision (TaTME) or abdominal transanal endoscopic microsurgery (TME) resections.
* Subjects must be Patients treated with curative intention.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Specific contraindications to laparoscopy.
* Intestinal obstruction or perforation.
* Histology other than adenocarcinoma.
* Subjects with rectal cancer arising in the background of inflammatory bowel disease.
* Subjects treated through local excision (ie, endoscopic, anorectal, or TEM approach).
* Subjects with synchronous metastases, except those with resectability criteria for the rectum.
* Subjects requiring a multivisceral resection or an abdominoperineal resection.
* Subjects converted to open technique.
* Subjects with history of fecal incontinence. Fecal incontinence (FI) will be defined based on Rome IV Criteria for Colorectal Disorders 31 as the uncontrolled passage of solid or liquid stool, occurring at least two times in a 4-week period.

Very low rectal cancers can cause a feeling of tenesmus associated with mucus leakage. As a result, patients will be asked if they had a bowel incontinence problem that dates back to a year ago (i.e. prior to the manifestation of current rectal cancer symptoms).

* Subjects with ultra-low rectal cancer where low anterior resection is converted to abdominoperineal resection intraoperatively due to sphincter involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men, women and members of all races and ethnic groups are eligible for this trial. Patients will be identified prospectively by the treating Co-Investigator surgeon according to the inclusion/exclusion criteria. The outpatient clinic schedule will be regularly screened ahead of time to identify potential candidates that fit the enrollment criteria.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
average change in anal resting pressure | Up to 6 months post-operation
  anal resting pressure will be estimated by taking measurements prior to operation and at 3-6 months post-operation. The mean change along with its 95% confidence interval will be reported for both groups
maximum squeeze pressure | Up to 6 months post-operation
  maximum squeeze pressure will be estimated by taking measurements prior to operation and at 3-6 months post-operation. The mean change along with its 95% confidence interval will be reported for both groups
Average intra-balloon pressure | Up to 6 months post-operation
  Average intra-balloon pressure will be estimated by taking measurements prior to operation and at 3-6 months post-operation. The mean change along with its 95% confidence interval will be reported for both groups

SECONDARY OUTCOMES:
Change in Fecal Incontinence Severity Index Score (FISI) | From before operation up to 12 weeks after operation
  Self-Reported, 4-question survey describing frequency of incontinence
Change in Cleveland Clinic Florida Fecal Incontinence (Wexner) score (CCF-FI) | From before operation up to 12 weeks after operation
  Self-Reported, 5-question survey scored 0-4 were higher scores indicate greater incontinence
Cleveland Clinic Global Quality of Life score (CGQL) | From before operation up to 12 weeks after operation
  Self-Reported, 4-question survey scored 1-10 where higher scores indicate greater quality of life
Low Anterior Resection Syndrome score (LARS) | From before operation up to 12 weeks after operation
  Self-Reported, 5-question survey with total scores ranging from 0-42 where higher scores indicating less bowel function

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Hull, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States